CLINICAL TRIAL: NCT04073576
Title: Randomized Cross Over Trial of the MiniMed™ 670G 4.0 Insulin Pump, Comparing Advanced Hybrid Closed Loop Mode With Sensor Augmented Pump Therapy in Type 1 Diabetes.
Brief Title: Assessment of Two Insulin Pump Insulin Delivery Systems in Type 1 Diabetes.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Christchurch Clinical Studies Trust Ltd (Industry)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CH-1803-AHCL
Record Dates: First submitted 2019-08-27; First posted 2019-08-29 (Actual); Last update posted 2019-08-29 (Actual); Status verified 2019-08

CONDITIONS: Type1diabetes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- AHCL (Experimental): Advanced Hybrid Closed Loop
  Interventions: Device: AHCL
- SAP+PLGM (Active Comparator): Sensor Augmented Pump with Predictive Low Glucose Monitoring
  Interventions: Device: SAP+PLGM

INTERVENTIONS:
Device: AHCL — Closed loop algorithm contained in the MiniMed™ 670G 4.0 pump to be used in the study; includes a modified proportional integrative derivative (PID) model, with insulin feedback, an auto correction bolus feature and additional safety features.
  Arms: AHCL
Device: SAP+PLGM — Sensor Augmented Pump (SAP) Therapy Mode with Predictive Low Glucose Management (PLGM), contained in the the MiniMed™ 670G 4.0 pump to be used in the study.
  Arms: SAP+PLGM

SUMMARY:
This is a study of the Minimed 670G 4.0 insulin pump, assessing the efficacy of the Advanced Hybrid Closed Loop (AHCL) algorithm in controlling blood glucose levels in Type 1 Diabetes.

DETAILED DESCRIPTION:
Insulin delivery systems are an increasingly popular treatment option for Type I Diabetes (T1D). Delivery systems consist of an insulin pump, a glucose sensor with a transmitter attached, and a maths program (algorithm) built into the pump. The algorithm uses sensor glucose levels to decide how much insulin should be delivered by the pump.

This study aims to see how well a new algorithm controls blood glucose levels in T1D. The study uses the MiniMed 670G 4.0 insulin pump and compares two different algorithms:

1. Advanced Hybrid Closed Loop (AHCL - the new algorithm)
2. Sensor augmented pump therapy with predictive low-glucose management (SAP with PLGM).

Approximately 60 participants with T1D, aged 7 - 80 years, will take part in the study.

Every participant will receive the following two treatment algorithms in random order, with a two-week washout between treatments:

* MiniMed 670G 4.0 insulin pump in AHCL mode for 4 weeks.
* MiniMed 670G 4.0 insulin pump in SAP + PLGM mode for 4 weeks.

During the study insulin pump data will be uploaded and changes in health will be monitored. In addition, participants will complete 3-day food diaries and a number of questionnaires. Participants at the Dunedin site will also be asked to complete home sleep studies during the trial (optional).

The results of the study will be used to further develop insulin delivery systems. It is hoped this may improve treatment for people with diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 7 - 80 years inclusive.
2. Type I diabetes as per the American Diabetes Association Classification, diagnosed at least 1 year prior to Study Day 1.
3. On insulin pump therapy for at least 6 months prior to study Day 1.
4. Minimum daily insulin requirement (Total Daily Dose) of greater than or equal to 8 units.
5. Willing and able to adhere to the study protocol.
6. Access to the internet and a computer system that meets requirements for uploading the study pump.

Exclusion Criteria:

1. Mean HbA1c more than 10.0% (86 mmol/mol) within 6 months prior to Study Day 1 (minimum of one test).
2. Use of a medication indicative of diabetes complications (ACE inhibitors and statins are permitted).
3. Use of systemic glucocorticoids within 2 weeks prior to the Baseline visit.
4. Current use of SGLT-2 or GLP-1 medications.
5. History or current evidence of significant seizure disorder, renal impairment or cardiovascular disease (including uncontrolled hypertension), in the opinion of the Investigator.
6. History of severe visual impairment, in the opinion of the Investigator.
7. If female, is pregnant or plans to become pregnant while participating in the study. A positive urine pregnancy test at Screening is exclusionary.
8. Any clinically significant concomitant disease or condition that could interfere with, or for which the treatment of might interfere with, the conduct of the study, or that would, in the opinion of the investigator, pose an unacceptable risk to the subject in this study.

Ages: 7 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-05-20 (Actual); Primary Completion 2019-10-11 (Estimated); Study Completion 2019-10-11 (Estimated)

PRIMARY OUTCOMES:
Performance of the AHCL system | 4 weeks
  percentage of sensor glucose values between 3.9 - 10.0 mmol/L

SECONDARY OUTCOMES:
Safety of the AHCL system | 4 weeks
  percentage of sensor glucose values <3.9 mmol/L and > 10 mmol/L

CONTACTS AND LOCATIONS:
Locations (1):
- Christchurch Clinical Studies Trust, Christchurch, Canterbury, New Zealand

IPD SHARING:
Plan to Share IPD: No